CLINICAL TRIAL: NCT00003538
Title: Stem Cell Augmented, Elutriated Grafts for Allogeneic Bone Marrow Transplantation
Brief Title: Prevention of Graft-Versus-Host Disease in Patients Undergoing Bone Marrow Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000066589, J9711; P30CA006973 (NIH); JHOC-97021903; JHOC-J9711; NCI-V98-1460
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Cancer
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent childhood acute lymphoblastic leukemia; recurrent adult Hodgkin lymphoma; recurrent childhood rhabdomyosarcoma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; Waldenstrom macroglobulinemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; myelodysplastic syndromes; Philadelphia chromosome positive chronic myelogenous leukemia; Philadelphia chromosome negative chronic myelogenous leukemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage II childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; recurrent ovarian germ cell tumor; chronic myelomonocytic leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV small lymphocytic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; anemia; graft versus host disease; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage I childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; non-Hodgkin lymphoma during pregnancy; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; childhood chronic myelogenous leukemia; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Neoplasms; Hodgkin Disease; Breast Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Carcinoma, Ovarian Epithelial; Neuroblastoma; Wilms Tumor; Waldenstrom Macroglobulinemia; Multiple Myeloma; Leukemia, Myeloid, Acute; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Hairy Cell; Recurrence; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Anemia; Graft vs Host Disease; Leukemia, Prolymphocytic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Therapeutics

INTERVENTIONS:
Biological: graft versus host disease prophylaxis/therapy
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: Bone marrow transplantation may be able to replace immune cells that were destroyed by chemotherapy or radiation therapy used to kill tumor cells. Sometimes the transplanted cells can make an immune response against the body's normal tissues. Stem cells that have been treated in the laboratory to remove lymphocytes may prevent this from happening.

PURPOSE: Clinical trial to prevent graft-versus-host disease in patients undergoing bone marrow transplantation.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether stem cell augmented, elutriated grafts prevent graft versus host disease in patients undergoing allogeneic bone marrow transplantation.

OUTLINE: Patients receive elutriated CD34+ augmented donor bone marrow on day 0.

Bone marrow samples are obtained before day 100, around 6 months, and 1 year after transplant.

PROJECTED ACCRUAL: Not specified

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one the following:

  * Acute myelogenous leukemia in CR1, ER1, CR2, ER2, CR3
  * Acute lymphocytic leukemia in CR1, ER1, CR2, ER2, CR3
  * Non-Hodgkin's lymphoma
  * Hodgkin's lymphoma
  * Multiple myeloma with no more than 12 months of prior alkylator based chemotherapy
  * Myelodysplastic syndrome (MDS)
  * Acute leukemia arising out of MDS
  * Primary resistant acute leukemia
  * Chronic myelomonocytic leukemia
  * Aplastic anemia (40 years of age and over)
  * Solid tumor malignancy (germ cell, sarcoma, breast, etc.)
  * Genetic disorders or inborn errors of metabolism as defined by preparative regimen protocol
  * Chronic myelogenous leukemia
* Must meet all inclusion criteria specified by the respective preparative regimen protocol
* No aplastic anemia under 40 years of age or myelofibrosis

PATIENT CHARACTERISTICS:

Age:

* 0.5 to 65

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior red blood cell or platelet transfusions from a sibling donor

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-03; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Jones, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] O'Donnell PV, Jones RJ, Vogelsang GB, Seber A, Ambinder RF, Flinn I, Miller C, Marcellus DC, Griffin C, Abrams R, Braine HG, Grever M, Hess AD, Piantadosi S, Noga SJ. CD34+ stem cell augmentation of elutriated allogeneic bone marrow grafts: results of a phase II clinical trial of engraftment and graft-versus-host disease prophylaxis in high-risk hematologic malignancies. Bone Marrow Transplant. 1998 Nov;22(10):947-55. doi: 10.1038/sj.bmt.1701476. PMID 9849691